CLINICAL TRIAL: NCT03586713
Title: Accuracy Of Sopro-Life Camera In Comparison With ICDAS II For Detection Of Initial Caries In Adult Patients With Non Cavitated Pits And Fissure Discoloration: Diagnostic Accuracy Study
Brief Title: Accuracy Of Sopro-Life Camera In Comparison With ICDAS II For Detection Of Initial Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura alzayyat, assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEBD-CU-2018-06-30
Record Dates: First submitted 2018-06-26; First posted 2018-07-16 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Screening of patients that come to the conservative dentistry department seeking dental care will continue until the target population is achieved. The patients' teeth will be subjected to visual examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the research investigator who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICDAS-II (Other): According to the international caries detection and assessment system (ICDAS-II). The visual examination was performed using the ICDAS-II criteria, which provides a standardized method of lesion detection. The ICDAS-II detection codes for coronal categories the score will be 0 =surface not restored or sealant then according to caries categories range from 0 to 6 depending on the severity of the lesion with the corresponding clinical views.
  Interventions: Diagnostic Test: light induced fluorescence camera

INTERVENTIONS:
Diagnostic Test: light induced fluorescence camera — The light induced fluorescence intraoral camera works with a visible blue light frequency (wavelength 450 nm) for the illumination of the dental surface and produces an overlapping image of the green fluorescence image on the image of the white light. The green fluorescence image is considered an indicator of healthy dental tissues. The colour of the fluorescence signal is green when the dentin is healthy. The healthy enamel is blue due to the scattered green light of the dentin, despite the lack of a fluorescence signal. On the other hand, caries can be easily detected by dark red fluorescence.

SUMMARY:
This study will be conducted to assess diagnostic predictive values of a light induced fluorescence intraoral camera versus those of the visual-tactile assessment method according to modified ICDAS-II criteria in clinical

DETAILED DESCRIPTION:
volunteers patients will be assigned in this study. Each patient should have at least one posterior tooth with pits and fissure discoloration and maximum 4 teeth. The teeth will be evaluated by two diagnostic methods (D), where D1 represents visual-tactile assessment method (ICDAS-II) and D2 represents light induced fluorescence intraoral camera.Three operators, the researcher and the 2 supervisors, from the Conservative Dentistry Department, Faculty of Dentistry, Cairo University, will be the examiners in this study. Each examiner will record the dental findings using both the visual- tactile assessment method and the fluorescent-aided identification method. The visual-tactile assessment method includes the use of mirror, probe under good illumination condition, while the fluorescent-aided identification method will be performed by light induced fluorescence intraoral camera.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 15 to 50 years.
* No gender restriction.
* Patients should have an acceptable oral hygiene level.
* Patients must have at least one posterior with fissure discoloration

Exclusion Criteria:

* • Patients with a compromised medical history.

  * Severe or active periodontal disease.
  * Heavy bruxism or a traumatic occlusion.
  * Acute or chronic dental infection.
  * Pregnant or breastfeeding women.
  * Patients with posterior restorations on molars or premolars.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
reliability and reproducibility of intra oral light fluorescence camera using kappa strength | 6 month
  in primary caries diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided